CLINICAL TRIAL: NCT05099848
Title: A Single-arm Exploratory Clinical Study of Conversion Treatment of Hepatic Arterial Infusion Chemotherapy Combined With Camrelizumab and Apatinib for Unresected Hepatocellular Carcinoma
Brief Title: A Trial of Conversion Treatment of HAIC Combined With Camrelizumab and Apatinib for Unresected Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Lei ZHAO, Doctor; Director, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-HCC-II-015
Record Dates: First submitted 2021-10-13; First posted 2021-10-29 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Camrelizumab; Apatinib; Hepatic artery infusion chemotherapy（HAIC）; Conversion therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab; apatinib; Folfox protocol; Oxaliplatin; Fluorouracil; Leucovorin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAHAIC group (Experimental): Hepatic Arterial Infusion Chemotherapy combined with Camrelizumab and Apatinib
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Procedure:
  1. Taking Apatinib-Mesylate Tablets (250 mg/tablet) orally on the 1st day 30minutes after meals, once a day, for continuous medication.
  2. On the 2nd day of treatment, intravenous infusion of Camrelizumab 200mg every 3 weeks.
  3. On the 3rd to 4th day of treatment, HAIC was conducted through a catheter intubated into the tumor feeding artery under DSA guidance with the following chemotherapeutic drugs (mFOLFOX, oxaliplatin 85 mg/m2 in 0-2 hours, folinic acid 400 mg/m2 in 2-3 hours, 5-FU 2500 mg/m2 46 hours) pumped into the tumor artery. The HAIC is repeated every 3 weeks. The cumulative maximum sessions of HAIC is up to 8 times.
  The cumulative maximum drug use period is up to 8 cycles. Patient will be administratied radical resection if possible during treatment. The patient is concurrent on medication until the treatment discontinuation criteria specified in the protocol appear.
  Other Names: Apatinib; FOLFOX Protocol (Oxaliplatin, fluorouracil, and leucovorin); Camrelizumab for injection and Apatinib-Mesylate Tablets

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of conversion treatment of Hepatic Arterial Infusion Chemotherapy combined with Camrelizumab and Apatinib for unresected hepatocellular carcinoma.

DETAILED DESCRIPTION:
A single-arm exploratory clinical study of conversion treatment of Hepatic Arterial Infusion Chemotherapy combined with Camrelizumab and Apatinib. After screening, subjects who meet the requirements for entry and exclusion signed the informed consent, received carrelizumab combined with apatinib and HAIC for conversion therapy, and After received 2-8 cycles (1 treatment cycle every 21 days) of HAIC combined camrelizumab and apatinib treatment, assess whether the subjects can undergo surgery every 2 cycles during the period: patients who are assessed as being able to undergo radical surgical resection receive elective radical resection surgery, and PD1 antibody should be stopped before surgery For 1 month, TKI drugs will be discontinued for 2-6 weeks; subjects who are assessed as not undergoing radical surgical resection will end this treatment plan. After leaving the group, they can receive any treatment according to the doctor's instructions and continue to follow up until the disease progresses and cannot be tolerated Toxic side effects, withdrawal of informed consent.

ELIGIBILITY:
Inclusion Criteria:

- 1. Subjects with hepatocellular carcinoma diagnosed or pathologically diagnosed according to the clinical diagnostic criteria of the diagnosis and treatment of primary liver cancer (2019 edition); 2. Subjects whose BCLC stage is B-C; 3. Subjects whose Child-Pugh is grade A; 4. Subjects whose the ECOG score is 0-1; 5. Subjects without extrahepatic metastases, no diffuse multiple tumors throughout the liver; 6. According to the researcher's assessment, subjects with hepatocellular carcinoma who do not have the conditions for radical resection, but are expected to achieve radical resection after conversion therapy, including but not limited to one of the following situations:

1. There are less than 3 tumors and mainly concentrated on the side of the liver;
2. Imaging proved to be combined with portal vein tumor thrombus (PVTT);
3. The investigator believes that other situations where radical resection may be achieved through conversion therapy.

7. Subjects whose estimated survival period is more than 3 months; 8. Subjects with at least one measurable lesion (according to the RECIST 1.1 standard, the long diameter of the CT scan of tumor lesions is ≥10mm, and the short diameter of CT scan of lymph node lesions is ≥15mm); 9. Newly treated subjects who have not undergone any local or systemic treatment for tumors in the past, and hepatocellular carcinoma patients who have undergone radical resection before recurrence after 2 years can be included; 10. Subjects' Routine laboratory tests (blood routine, liver and kidney function, coagulation function, etc.) have no significant abnormalities 11. Subjects with potential for childbirth need to use a medically approved contraceptive method (such as intrauterine device, contraceptive pill or condom) during the study treatment period and within 1 month after the end of the study treatment period; and The serum or urine HCG test within 72 hours before study entry must be negative, and it must be a non-lactating period; 12.18-80 years old; 13. Subjects participated in the study voluntarily, without mental illness or other mental symptoms, with full civil capacity, signed informed consent, good compliance, and able to cooperate with follow-up.

Exclusion Criteria:

- 1. Previously diagnosed by histology/cytology with fibrous lamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma and other components; 2. A history of hepatic encephalopathy, or a history of liver transplantation; 3. A history of allergies to test drugs: Camrelizumab and any component of other drugs; 4. The subject's refractory pleural or pericardial effusion is poorly controlled; 5. Previously received anti-PD-1 or PD-L1 or CTLA-4 or Car-T immunotherapy; 6. Except for history of interstitial lung disease (radiation pneumonia that has not been treated with hormones), history of non-infectious pneumonia; 7. The subject has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis , Nephritis, hyperthyroidism, reduced thyroid function; subjects suffering from vitiligo or asthma in childhood has completely resolved, and no intervention after adults can be included; subjects with asthma requiring bronchodilators for medical intervention can not be included ); 8. The subject is using immunosuppressive agents, or systemic or absorbable local hormone therapy to achieve immunosuppressive purposes (dose>10mg/day prednisone or other curative hormones), and within 2 weeks before enrollment Still in use; 9. Severe infections (CTCAE> level 2) occurred 4 weeks before the first use of the study drug; 10. The subject has experienced acute cardiovascular and cerebrovascular diseases such as acute cerebral infarction, acute coronary syndrome, etc. and the cardiovascular clinical symptoms or diseases within one month are not well controlled; 11. According to NYHA standards, grade Ⅲ to Ⅳ cardiac insufficiency, or cardiac color Doppler ultrasound examination reveals that the left ventricular ejection fraction (LVEF) is less than 50%; 12. Patients with a clear gastrointestinal bleeding tendency, including the following conditions: local active ulcer lesions, and fecal occult blood {(＋＋) can not be included in the group}; patients with a history of melena and hematemesis within 2 months; 13. Abnormal blood coagulation function (INR>1.5APTT>1.5ULN), with bleeding tendency; 14. Long-term unhealed wounds or fractures; major surgical operations or severe traumatic injuries, fractures or ulcers occurred within 4 weeks; 15. Subjects with congenital or acquired immune deficiencies (such as HIV infection), or active hepatitis (hepatitis B reference: HBV DNA test value exceeding 2000 IU/ml) need to be excluded; if the patient has active hepatitis B virus (HBV) infection: HBV-deoxyribonucleic acid (DNA<2000 IU/mL, and received anti-HBV therapy for at least 14 days before randomization and is willing to receive antiviral therapy throughout the study period (recommended nucleoside analogs, such as entecavir or alternative Norfovir dipivoxil, etc.) can be included in the study.

16. Patients with a history of psychotropic drug abuse and unable to quit or patients with mental disorders; 17. According to the judgment of the investigator, patients with concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study; 18. The researcher believes that it is not suitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | within 28 working days after operation
  the complete resection rate of all tumor under microscope
Surgical conversion rate | within 28 working days after operation
  Surgical conversion rate was defined as the proportion of subjects with successful conversion over all subjects who received conversion treatment

SECONDARY OUTCOMES:
MPR | within 14 working days after operation
  MPR rate was defined as the percentage of patients who achieved a major pathological response (residual tumor ≤10%)
Objective response rate (ORR) by RECIST 1.1 and mRECIST | From date of first dose of study drug until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to approximately 3 years)
  ORR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by RECIST 1.1 and mRECIST
The disease control rate (DCR) | From date of first dose of study drug until disease progression, stable disease, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to approximately 3 years)
  DCR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) or stable disease (SD) at the time of data cutoff as assessed by RECIST 1.1 and mRECIST
Duration of response (DOR) by RECIST 1.1 and mRECIST | From the first documentation of CR or PR to the first date of documentation of disease progression or death whichever occurs first (up to approximately 3 years)
  DOR is defined as the time from the first documentation of CR or PR to the date of first documentation of disease progression or death (whichever occurs first) as assessed by RECIST 1.1 and mRECIST
The progression-free survival time (PFS) | From the first documentation of PD to the first date of documentation of disease progression or death whichever occurs first (up to approximately 3 years)
  The progression-free survival time (PFS) defined as the time from the first study dose date to the date of first documentation of disease progression as assessed by RECIST 1.1 and mRECIST
The overall survival time (OS) | Up to ~4 years
  OS is measured from the start date of the Treatment Phase (date of first study dose) until date of death from any cause.
The overall survival rate of 1-year and 2-year(1-year and 2-year OSR) | From date of first dose of study drug to the date of first documentation of death from any cause, whichever occurs first (up to approximately 3 years)
  Up to ~3 years
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to ~1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhao, MD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yalikun K, Li Z, Zhang J, Chang Z, Li M, Sun Z, Liu Z, Yang Y, Xu L, Li L, Zhang C, Sun P, Zhong J, Cui K, Shi X, Zhang B, Zhao L. Hepatic artery infusion chemotherapy combined with camrelizumab and apatinib as conversion therapy for patients with unresectable hepatocellular carcinoma: a single-arm exploratory trial. BMC Cancer. 2025 May 7;25(1):838. doi: 10.1186/s12885-025-14250-5. PMID 40335980